CLINICAL TRIAL: NCT06207552
Title: A Single-arm, Open Label, Single-dose Clinical Study to Evaluate the Safety, Tolerability and Efficacy of BBM-F101 Injection in the Treatment of Pediatric Fabry Disease
Brief Title: Evaluation of the Safety, Tolerability and Efficacy of a Gene Therapy Drug for the Treatment of Pediatric Fabry Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM017-IIT1001
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Fabry Disease
Keywords: Fabry
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of BBM-F101 injection (Experimental): The dose of BBM-F101 injection will be calculated according to the participant's weight with single intravenous infusion.
  Interventions: Genetic: BBM-F101 injection

INTERVENTIONS:
Genetic: BBM-F101 injection — The dose of BBM-F101 injection will be calculated according to the participant's weight with single intravenous infusion.

SUMMARY:
This is a single-arm, open label, single-dose clinical study to evaluate the safety, tolerability and efficacy of BBM-F101 injection in the pediatric Fabry disease participants up to 52 weeks after infusion, and the long-term safety and efficacy of BBM-F101 injection up to 5 years after infusion.

BBM-F101 injection is an adeno-associated virus (AAV) gene therapy product for the treatment of pediatric Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

1. The participant's legal guardian fully understands the objectives, nature, methods and potential risks of the study and signs a written informed consent; If the participant is >= 8 years old, the participant must also agree to participate in the study and sign a written informed consent;
2. Decreased α-Gal A (α-galactosidase A) and confirmed diagnosis of Fabry Disease by genetic testing;
3. Males or females aged ≥7 years and <18 years old;
4. Acceptable eGFR (estimated Glomerular Filtration Rate) result in screening period;
5. Participants had at least one of the clinical manifestations for Fabry disease;
6. Acceptable capsid antibody titers;
7. Acceptable anti α-Gal A antibody titers;
8. Acceptable laboratory values;
9. Participant's legal guardian and participant with good cooperation and compliance;
10. Use of reliable contraception methods during the study for adolescence.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B virus DNA (HBV-DNA), positive for hepatitis C virus RNA (HCV-RNA), positive for HIV or syphilis;
2. Have potential liver diseases;
3. Heart failure and severe arrhythmias;
4. Severe allergic reactions for enzyme replacement drugs or other medications;
5. Acute/chronic infections;
6. End-stage renal disease;
7. Have a vaccination history within 30 days prior to screening, or have a vaccination plan during the screening period and the main study period;
8. Have received gene therapy or used other investigational drugs within four weeks prior to dosing;
9. Other conditions that make the participant not eligible for the study according to the investigator.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limited toxicity | 12 weeks
  The incidence of dose limited toxicity (DLT) events as determined by the safety review committee (SRC) within DLT observation period following the BBM-F101 injection
Incidence of adverse events and serious adverse events | 52 weeks
  The incidence of adverse events (AE) and serious adverse events (SAE) within 52 weeks following the BBM-F101 injection

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, MD,PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No